CLINICAL TRIAL: NCT01235182
Title: Combination of Lung Ultrasound(a Comet-tail Sign) and N-terminal Pro-brain Natriuretic Paptide in Differentiating Acute Dyspnea in Prehospital Emergency Setting
Brief Title: Ultrasound in Acute Dyspnea in the Field
Status: Completed | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Prof.Štefek Grmec, MD,PhD, Zdravstveni dom Adolfa Drolca Maribor, Center for Emergency Medicine Maribor
Other Study IDs: ADMB2010
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2007-07

CONDITIONS: Heart Failure; COPD; Asthma
Keywords: acute dyspnea; prehospital emergency setting; differential diagnosis; ultrasound; NT-proBNP
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute dyspnea, field, diagnostic: All patients with shortness of breath as the primary complaint (defined as eitherthe sudden onset of dyspnea without history of chronic dyspnea or an increase in the severity of chronic dyspnea and were age >18 years.

SUMMARY:
Acute heart failure is one of the main causes of acute respiratory distres in prehospital emergency setting. The early and correct diagnosis is important because the misdiagnosis can result in deleterious consequeance to patients. Rapid bedside tests (like NT-proBNP) and point-of-care lung ultrasound could be useful methods in field. This study confirmed that the combination of ultrasound sign in combination with rapid NT-proBNP test has a hibh diagnostic accuracy in differentiating between cardiac and pulmonray causes of acute dyspnea in the field and the tretament possibilities in clinical obscure cases are mainly improved.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criterion for the study was shortness of breath as the primary complaint (defined as either the sudden onset of dyspnea without history of chronic dyspnea or an increase in the severity of chronic dyspnea).

Exclusion Criteria:

* Exclusion criteria were age <18 years, history of renal insufficiency, trauma, severe coronary ischemia (unless patient's predominant presentation was dyspnea), and other causes of dyspnea: pneumonia, pulmonary embolism, carcinoma, pneumothorax, pleural effusion, intoxications (drugs), anaphylactic reactions, upper airway obstruction, bronchial stenosis, and gastroesophageal reflux disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute dyspnea in the time o the investigation in the field-prehospital settingInclusion criterion for the study was shortness of breath as the primary complaint (defined as either the sudden onset of dyspnea without history of chronic dyspnea or an increase in the severity of chronic dyspnea). Exclusion criteria were age <18 years, history of renal insufficiency, trauma, severe coronary ischemia (unless patient's predominant presentation was dyspnea), and other causes of dyspnea: pneumonia, pulmonary embolism, carcinoma, pneumothorax, pleural effusion, intoxications (drugs), anaphylactic reactions, upper airway obstruction, bronchial stenosis, and gastroesophageal reflux disorder, according to the history, clinical status, and additional laboratory tests available in prehospital setting (D-dimer, troponin, C-reactive protein)
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Štefek Grmec, MD,PhD,Prof., Principal Investigator — Center of Health Center for Emergency Medicine Maribor
Locations (1):
- Center for Emergency Medicine maribor, Maribor, Slovenia

REFERENCES:
- [Background] Klemen P, Golub M, Grmec S. Combination of quantitative capnometry, N-terminal pro-brain natriuretic peptide, and clinical assessment in differentiating acute heart failure from pulmonary disease as cause of acute dyspnea in pre-hospital emergency setting: study of diagnostic accuracy. Croat Med J. 2009 Apr;50(2):133-42. doi: 10.3325/cmj.2009.50.133. PMID 19399946
- [Derived] Prosen G, Klemen P, Strnad M, Grmec S. Combination of lung ultrasound (a comet-tail sign) and N-terminal pro-brain natriuretic peptide in differentiating acute heart failure from chronic obstructive pulmonary disease and asthma as cause of acute dyspnea in prehospital emergency setting. Crit Care. 2011;15(2):R114. doi: 10.1186/cc10140. Epub 2011 Apr 14. PMID 21492424